CLINICAL TRIAL: NCT02843711
Title: Molecular Analysis of 150 Lung Adenocarcinoma With Corresponding Histopathological and Clinical Data Available
Brief Title: Molecular Analysis of 150 Lung Adenocarcinoma
Acronym: LUNG-EST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0161
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Lung Adenocarcinoma
Keywords: Lungcarta Panel; lung adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paraffin-embedded formalin fixed tumour sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adenocarcinoma: Tumour samples coming from patients harboring a lung adenocarcinoma diagnosed at the Hospices Civils de Lyon. Tumour samples are coming from lung surgery.
  Interventions: Genetic: Sequencing

INTERVENTIONS:
Genetic: Sequencing — Tumour samples are coming from routine histopathological procedure. They are used with consent of the patients. Genomic DNA extraction is performed from paraffin-embedded formalin-fixed (FFPE) tumour samples of lung adenocarcinoma. The genomic DNA mutations are identified by mass spectrometry array (Sequenom) using the LungCarta Panel. This panel could identify 214 mutations among 26 oncogenes.

SUMMARY:
LUNG-EST is a retrospective study including 152 patients who benefit from lung surgery during the years 2012 to 2013 at Hospices civils de Lyon and with a diagnosis of lung adenocarcinomas. For all patients, clinical data and histopathological data are available. The objective of this study is to characterize these lung adenocarcinomas by the LungCarta Panel using the mass spectrometry array Sequenom. This panel could identify 214 DNA mutations and/or frameshift insert/deletion among 26 oncogenes. Once included in the study, the adenocarcinomas are also included in a Tissue MicroArray (TMA) in order to perform immunohistochemical analysis. Immunohistochemical staining with innovative antibodies are correlated with clinical, histopathological and molecular data.

Our hypothesis is that this TMA could constitute a good tool to screen interesting protein's expression.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* lung adenocarcinoma
* Surgical specimen

Exclusion Criteria:

* not adenocarcinoma subtype of lung cancer
* Tumour biopsy
* insufficient material for DNA extraction

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults>18 years old with diagnosis of lung adenocarcinoma and treatment by surgery
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Genomic DNA Mutation | at diagnosis (Day 0)
  Mutations identified by the LungCarta Panel (Sequenom) at the time of diagnosis. DNA was extracted from the lung surgical specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Marie BREVET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Anatomie et cytologie pathologiques Groupement hospitalier Est, Institut de cancérologie des Hospices civils de Lyon,, Lyon, France